CLINICAL TRIAL: NCT05282706
Title: A Placebo-controlled Clinical Trial Investigating the Use of Aromatherapy in Conjunction With Physical/Occupational Therapy in an Acute Care Setting
Brief Title: Use of Aromatherapy in Conjunction With Physical/Occupational Therapy in an Acute Care Setting
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: University Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC20210769H
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Suffering, Physical; Nausea
Keywords: Acute Care; Physical Therapy; Occupational Therapy; Aromatherapy
MeSH Terms: conditions — Pain; Nausea | interventions — lavender oil; peppermint oil

STUDY DESIGN:
Intervention Model Description: Three interventional and one control arm
Who Masked: Participant
Masking Description: Subjects will be assigned to an arm based upon the symptoms they are experiencing prior to their therapy session. If a patient reports nausea symptom, they will be assigned to the peppermint fragrance or a placebo. The randomization will be conducted in a 1:2 ratio, one placebo to two experimental. If a patient reports pain symptom, they will be assigned to the lavender or mandarin fragrance or placebo. The randomization will be conducted in a 1:2 ratio, one placebo to two experimental. The experimental group will then be randomized to a 1:1 ratio between lavender and mandarin. For those that refuse the aromatherapy patch will be asked to serve as a control and receive usual care with no patch.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Pain Symptoms Arm (Experimental): Subjects who will receive physical or occupational therapy experiencing pain prior to therapy session.
  Interventions: Drug: Lavender Oil; Drug: Mandarin Oil
- Nausea Symptom Arm (Experimental): Subjects who will receive physical or occupational therapy experiencing nausea prior to therapy session.
  Interventions: Drug: Peppermint oil
- Placebo Group (Placebo Comparator): Subjects who will receive physical or occupational therapy experiencing pain or nausea prior to therapy session.
  Interventions: Other: Placebo
- Standard of Care Group (No Intervention): Subjects who will receive physical or occupational therapy experiencing pain or nausea prior to therapy session that decline the option to use an aromatherapy patch.

INTERVENTIONS:
Drug: Lavender Oil — A hydrogel lavender oil infused aromatherapy patch
  Other Names: Lavender Aromatherapy Patch
  Arms: Pain Symptoms Arm
Drug: Mandarin Oil — A hydrogel mandarin oil infused aromatherapy patch
  Other Names: Mandarin Aromatherapy Patch
  Arms: Pain Symptoms Arm
Drug: Peppermint oil — A hydrogel peppermint oil infused aromatherapy patch
  Other Names: Peppermint Aromatherapy Patch
  Arms: Nausea Symptom Arm
Other: Placebo — A placebo patch containing no aromatherapy oil
  Other Names: Placebo patch
  Arms: Placebo Group

SUMMARY:
Use of inhaled essential oils to reduce the symptoms of pain or nausea, enabling a patient to have increase participation with PT or OT, thereby minimizing hospitalization-related risks and potentially reducing the length of stay in the hospital.

DETAILED DESCRIPTION:
The study intervention consists of 3 essential oils: lavender, mandarin and peppermint administered on an inhalation patch affixed in the chest region of the participant gown. The inhalation patch consists of hydrogel cast onto polyester film, supported by non-woven polyester fabric, covered with a polyethylene film. The proprietary foil-backed lamination on the patch is used to provide an occlusive barrier that prevents any essential oil from being absorbed through the skin. The placebo will consist of a comparable sized felt patch with adhesive backing with no essential oil applied.

ELIGIBILITY:
Inclusion Criteria:

1. Inpatients of acute care setting at University Health hospital
2. Provision of a signed and dated informed consent form
3. English or Spanish speaking
4. Male or Female, aged 18 years and older
5. Willing to comply with all study procedures

Exclusion Criteria:

1. Respiratory disorders, e.g., asthma, chronic obstructive pulmonary disease (COPD), chronic bronchitis, emphysema, lung cancer, cystic fibrosis, pneumonia, pleural effusion
2. Cognitive impairment
3. Unable to communicate
4. Admitted to the closed access unit or to psychiatry
5. Allergic to lavender, mandarin or peppermint oil
6. Diseases that cause olfactory disorders such as: COVID-19, benign growths or polyps, congestion from a cold, sinus infection or allergy flare-up
7. Drugs that may cause loss of the ability to smell e.g., intranasal zinc products, decongestant nose sprays and certain oral drugs such as nifedipine and phenothiazines
8. Pregnant women (self-reported)
9. Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Completion of PT/OT session | 30 minutes
  The number of subjects who successfully completed physical or occupational therapy session

SECONDARY OUTCOMES:
Change in Pain/Nausea Scale | Baseline to post therapy follow-up (30 minutes)
  A scale with ranks the pain or nausea from 0 to 10 with a 0 being no pain or nausea and 10 being the worst pain

OTHER OUTCOMES:
Increase in participation in PT and OT sessions | 30 minutes
  An exploratory measure to compare whether the use of aromatherapy changes the number of participants in PT or OT.

CONTACTS AND LOCATIONS:
Overall Officials: Bianca Gonzales, OTR, CNT, EdD, MOT, Principal Investigator — University Health
Locations (1):
- Bianca Gonzales, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The study will be registered on ClinicalTrials.gov and will be conducted in accordance with the ICMJE publication and data sharing policies and regulations.
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available once analyzed and published